CLINICAL TRIAL: NCT06649643
Title: Inbon Errors of Immunity Attending Assiut University Children&Amp;#39;s Hospital: a Single Center Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christeena Goda Hakeem, Inbon errors of immunity attending Assiut University Children's Hospital: a single center study, Assiut University
Other Study IDs: IEIs of Assuit hospital
Record Dates: First submitted 2024-09-27; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Inborn errors of immunity — A. Routine
  .1CBC with blood film.
  .2Liver Function Test.
  .3Kidney Function Test.
  4. Inflamatory marker ESR, CRP
  B.Immunology
  1. Immunoglobulins IgG, IgM, IgA, IgE
  2. Flow cytometric assessment: B Cell (CD19), T cells (CD3,CD4, CD8) anc NK Cells (CD16+56) and other markers whenever needed (e.g. CD40, CD40L for cases of hyper IGM)
  3. Chest x-ray to assess thymus and any abnormality
  4. DHR123 whenever needed (e.g. chronic granulomatous disease).
  5. LAD panel (CD11b CD15-CD18) whenever needed.
  6. Complement assay (CH
Diagnostic Test: A. Routine .1CBC with blood film. .2Liver Function Test. .3Kidney Function Test. 4. Inflamatory marker ESR, CRP B.Immunology 1-Immunoglobulins IgG, IgM, IgA, IgE 2-Flow cytometric assessment: B — A. Routine
  .1CBC with blood film.
  .2Liver Function Test.
  .3Kidney Function Test.
  4. Inflamatory marker ESR, CRP
  B.Immunology
  1. Immunoglobulins IgG, IgM, IgA, IgE
  2. Flow cytometric assessment: B Cell (CD19), T cells (CD3,CD4, CD8) anc NK Cells (CD16+56) and other markers whenever needed (e.g. CD40, CD40L for cases of hyper IGM)
  3. Chest x-ray to assess thymus and any abnormality
  4. DHR123 whenever needed (e.g. chronic granulomatous disease).
  5. LAD panel (CD11b CD15-CD18) whenever needed.
  6. Complement assay (CH

SUMMARY:
Aim of Study The aim of this study to describe the clinical profile of children diagnosed as IEIs who were admitted to in Assiut university children's Hospital.

DETAILED DESCRIPTION:
Introduction

Inborn errors of immunity (IEIs) are generally considered to be rare monogenic disorders of the immune system that cause immunodeficiency, autoinflammation, autoimmunity, allergy and/or cancer (1). IEIs are a group of diseases comprised of more than 450 IEIs, and they are becoming more prevalent (2). Although IEIs are rare diseases, they are more common than previously thought, following the use of modern diagnostic methods. A recent evaluation indicated that at least 1-2% of the world's population are affected by IEIs (3). Several warning signs have been developed to increase physician awareness about the early signs that can help to diagnosis IEIs. Warning signs of IEIs were developed by an institution called the Jeffrey Modell Foundation (JMF) (4,5). the ten warning signs are four or more new ear infections within 1 year,two or more serious sinus infections within 1 year,two or more months on antibiotics with little effect,two or more pneumonias within 1 year,failure of an infant to gain weight or grow normally,recurrent, deep skin or organ abscesses, persistent thrush in mouth or fungal infection on skin, need for intravenous antibiotics to clear infections,Two or more deep-seated infections including septicemia and family history of IEIs. (6). The International Union of Immunological Societies (IUIS) has classified IEIs into nine categories based upon the segment of the immune system that is affected, plus a 10th category of IEIs phenocopies. Each category is characterized by unique types of infections and clinical features that are useful for the selection of initial appropriate laboratory evaluation to help with diagnosis (7). The mechanisms that explain the increased susceptibility of IEIs patients to the development of tumours are multiple and different in the various pathologies. The most common process is the reduction of cell-mediated immunosurveillance, which plays a fundamental role in protecting against tumours (8,9). Several pathways, such as genomic instability, overstimulation of immune cells, viral infection and chronic inflammation, have been proposed to explain the increased incidence of malignancy among patients with IEIs (10). Moreover, defective dendritic cells (DCs) differentiation and function, which affect the initiation and development of T cell responses, have been associated with cancer development (11) The diagnostic investigation of IEIs should be guided by the clinical characterization of patients, aiming to optimize the use of complementary tests. Many diagnoses are attained only through genetic tests, which are not always available. However, the absence of a diagnosis of certainty should never delay the implementation of therapeutic measures that preserve patient life and health (12). Major advances in the treatment of these disorders have occurred over the last half-century, and deeper molecular understanding of many disorders combined with clinically available genetic testing is allowing for use of precision therapy for several IEIs. Patients with antibody deficiencies who rely on immunoglobulin replacement therapy now have many treatment options with products that are much safer and better tolerated compared to the past (13). Steroids are often used as an initial therapy but have serious long-term complications. Targeted immune therapies, such as cytokine or small molecule inhibitors, are increasingly available with the advantage of fewer global immune suppressive effects. However, patients with IEIs often do not have an adequate clinical response to immunosuppressive treatment, resulting in referral for allogeneic hematopoietic cell transplantation (HCT) as a potentially curative therapy (14,15).

ELIGIBILITY:
Inclusion Criteria:patients with the ten warning signs are four or more new ear

infections within 1 year,two or more serious sinus infections within 1 year,two or more months on antibiotics with little effect,two or more pneumonias within 1 year,failure of an infant to gain weight or grow normally,recurrent, deep skin or organ abscesses, persistent thrush in mouth or fungal infection on skin, need for intravenous antibiotics to clear infections,Two or more deep-seated infections including septicemia and family history of IEIs -

Exclusion Criteria:

* patients without any criteria of ten warning signs

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sex- all Age - maximum age 18 y
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Profile of Patients with Inborn Errors of Immunity in Assiut University Children Hospital: Single Center Study | Baseline
  Warning signs for early diagnosis
  * Weight in kilogram
  * Height in meters investigation
    --Routine
  * CBC with blood film.
  * Liver Function Test.
  * Kidney Function Test.
  * Inflammatory marker ESR,CRP
    --Immunology
  * Immunoglobulins IgG, IgM, IgA, IgE
  * Flow cytometric assessment: B Cell (CD19), T cells (CD3,CD4, CD8) and NK Cells (CD16+56) and other markers whenever needed (e.g. CD40, CD40L for cases of hyper IGM)
  * Chest x-ray to assess thymus and any abnormality
  * DHR123 whenever needed (e.g. chronic granulomatous disease).
  * LAD panel ( CD11b CD15- CD18) whenever needed. .Complement assay (CH 50,C3,C4) whenever needed .

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tangye SG, Al-Herz W, Bousfiha A, Chatila T, Cunningham-Rundles C, Etzioni A, Franco JL, Holland SM, Klein C, Morio T, Ochs HD, Oksenhendler E, Picard C, Puck J, Torgerson TR, Casanova JL, Sullivan KE. Correction to: Human Inborn Errors of Immunity: 2019 Update on the Classification from the International Union of Immunological Societies Expert Committee. J Clin Immunol. 2020 Jan;40(1):65. doi: 10.1007/s10875-020-00763-0. PMID 32086639
- [Result] Tangye SG, Al-Herz W, Bousfiha A, Cunningham-Rundles C, Franco JL, Holland SM, Klein C, Morio T, Oksenhendler E, Picard C, Puel A, Puck J, Seppanen MRJ, Somech R, Su HC, Sullivan KE, Torgerson TR, Meyts I. Human Inborn Errors of Immunity: 2022 Update on the Classification from the International Union of Immunological Societies Expert Committee. J Clin Immunol. 2022 Oct;42(7):1473-1507. doi: 10.1007/s10875-022-01289-3. Epub 2022 Jun 24. PMID 35748970